CLINICAL TRIAL: NCT01014507
Title: Randomisierte Phase II Studie Zum Einsatz Von Goserelin Und Oralen Kontrazeptiva Zur Reduktion Ovarieller Toxizitäten während Zytostatischer Primärtherapie Bei Fertilen Patientinnen Mit Hodgkin Lymphom in Fortgeschrittenen Stadien
Brief Title: Protection of Ovarian Function in Female Patients With Hodgkin Lymphoma
Acronym: PROFE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: German Hodgkin Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROFE
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2011-10

CONDITIONS: Hodgkins Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Contraceptives, Oral; Goserelin

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: 8 cycles BEACOPPesc plus oral contraceptive
- B (Experimental)
  Interventions: Drug: 8 cycles BEACOPPesc plus Goserelin

INTERVENTIONS:
Drug: 8 cycles BEACOPPesc plus oral contraceptive
  Arms: A
Drug: 8 cycles BEACOPPesc plus Goserelin
  Arms: B

SUMMARY:
This study is designed to test the the protective capacity of Goserelin compared with oral contraceptive

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage Hodgkins Lymphoma (histologically proven)
* Normal FSH-levels
* Written informed consent

Exclusion Criteria:

* Hodgkins Lymphoma as "composite lymphoma"
* Primary ovarial dysfunction
* Age > 40

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2004-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
FSH level 6 month after end of treatment | 6 month

REFERENCES:
- [Result] Behringer K, Wildt L, Mueller H, Mattle V, Ganitis P, van den Hoonaard B, Ott HW, Hofer S, Pluetschow A, Diehl V, Engert A, Borchmann P; German Hodgkin Study Group. No protection of the ovarian follicle pool with the use of GnRH-analogues or oral contraceptives in young women treated with escalated BEACOPP for advanced-stage Hodgkin lymphoma. Final results of a phase II trial from the German Hodgkin Study Group. Ann Oncol. 2010 Oct;21(10):2052-2060. doi: 10.1093/annonc/mdq066. Epub 2010 Mar 19. PMID 20305034